CLINICAL TRIAL: NCT04135027
Title: Study of Factors and Mechanisms Influencing the Effects of Treatments in Crohn's Disease Patients (a Prospective, Observational Cohort Designed for Precise Evaluation, Personalized RIsk Stratification and Targeted Treatment (PRIST Cohort))
Brief Title: Study of Factors and Mechanisms Influencing the Effects of Treatments in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IR2019001055
Record Dates: First submitted 2019-10-02; First posted 2019-10-22 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cell(PBMCs) were collected from patients and volunteers using Ficoll-PaqueTM PLUS medium (GE Healthcare, Uppsala, Sweden), and total RNA was extracted using TRIzol reagent (Ambion, Carlsbad, CA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CD group: no interventions
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
The course of Crohn's disease (CD) varies considerably between patients, but reliable prognostic markers are not available in clinical practice. Even though several parameters have been associated with prognosis in CD-including clinical features, serology and genetic variants-none are sufficient to guide therapy in clinical practice. Trying to find out the mechanisms influencing the effectiveness of treatments and develop a personalized therapy is an urgent problem in the era of biologics as the investigators now have a growing armamentarium of IBD therapies. Several scientists found that the levels of T cells subsets ratio and inflammation cytokines were significantly increased in the intestinal mucosa and serum in active IBD patients, whereas mucosal innate lymph cells had specific effects in inflammation. However the studies about the differences of lymph cell levels between subgroups of IBD patients and their relationships with effectiveness of treatments are relatively rare. Based on above, the investigators plan to recruit patients diagnosed and suspicious of Crohn's disease and a group of diseases in differential diagnosis of CD to keep track of their disease characteristics, therapy and response, collect their blood sample at specific points of time, to investigate the mechanisms of heterogeneity of therapy effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or Previously diagnosed of Crohn's disease according to 2010 WGO criteria for Crohn's disease
* Aged 14-80 years old.

Exclusion Criteria:

* History of malignancy
* Pregnant/breastfeeding at screening
* Other serious medical or psychiatric illness.
* Unable to comply with protocol requirements

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 14-80 years old, newly diagnosed or previously diagnosed of Crohn's disease according to 2010 WGO criteria for Crohn's disease were recruited from a specialist IBD clinic.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
time to first treatment escalation | 6 months to 1 year
  time to first treatment escalation
bowel surgery | 1 month to 1 year
  time to receive bowel surgery after diagnosis

SECONDARY OUTCOMES:
side effects of medications | 1 month to 1 year
  side effects of medications including infection and malignancy etc.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Chongqing Hospital of the University of Chinese Academy of Sciences (Chongqing People's Hospital), Chongqing, Chongqing Municipality
  - Nanjing Drum Tower Hospital (Nanjing Gulou Yi Yuan), the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - 2nd Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang
  - Huadong Hospital affiliated to Fudan University, Shanghai